CLINICAL TRIAL: NCT05060471
Title: Neoadjuvant PD-1 Blockade Combined with Chemotherapy Followed by Concurrent Immunoradiotherapy for Locally Advanced Anal Canal Squamous Carcinoma Patients
Brief Title: PD-1 Blockade Combined with Chemotherapy Followed by Concurrent Immunoradiotherapy for Locally Advanced SCCA Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yuan-hong Gao, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2021-137-01
Record Dates: First submitted 2021-09-19; First posted 2021-09-29 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Anal Canal Cancer; Anal Squamous Cell Carcinoma; Anal Cancer; Anal Canal Cancer Stage I; Anal Canal Cancer Stage II; Anal Canal Cancer Stage III
MeSH Terms: conditions — Anal Canal Carcinoma; Anus Neoplasms | interventions — toripalimab; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervetional group (Experimental): Neoadjuvant PD-1 antibody toripalimab combined with docetaxol and cisplatin, followed by radiotherapy and concurrent toripalimab
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab — Four cycles of neoadjuvant PD-1 antibody toripalimab combined with docetaxol and cisplatin, followed by radiotherapy and two cycles of concurrent toripalimab.
  Other Names: radiation

SUMMARY:
Locally Advanced Anal Canal Squamous Carcinoma Patients will be enrolled and given four cycles of neoadjuvant PD-1 antibody toripalimab combined with docetaxol and cisplatin, followed by radiotherapy and two cycles of concurrent toripalimab. Treatment outcomes and toxicities will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

(1) Histology confirmed as anal canal squamous carcinoma;

1. Clinical stage I-III
2. No distant metastasis;
3. Age: 18-75 years old;
4. ECOG 0-1 score
5. Adequate bone marrow, liver, kidney function
6. if HIV infected, HIV loading is below the lower limit (<20 copy </ ml), with the number of CD4+T cells > 300> ml
7. Non-pregnant or lactating women;
8. No other malignant disease within 5 years before diagnosis of anal cancer squamous carcinoma (except endocervical cancer in situ or skin basal cell carcinoma which had been cured); no other malignant disease beside anal cancer squamous carcinoma
9. No other serious disease leading to shortened survival.
10. No previous anal canal surgery or anal tumor resection (except for biopsy);
11. No chemotherapy received within the previous 5 years;
12. No previous pelvic radiation;
13. No biological treatment received in the previous 5 years;
14. No previous immunotherapy received.

Exclusion Criteria:

1. Diagnosed as stage I and well differentiated squamous cell carcinoma
2. Distant metastasis
3. Received radiation therapy in abdominal or pelvic regions
4. Pregnant, lactating woman patient or fertile but lacks adequate contraceptives
5. Infectious disease: Active phase chronic hepatitis B or hepatitis C (high copies of virus DNA); Other serious active clinical infection
6. Patients with active tuberculosis (TB) are receiving anti-tuberculosis treatment or have received anti-tuberculosis treatment within 1 year before screening;
7. Chronic inflammatory colorectal disease, unrelieved ileus
8. Dyscrasia or organ decompensation
9. Allergic to research-related drugs
10. Severe hypertension with poor drug control;
11. Epilepsy require medical treatment (such as steroid or antiepileptic therapy);
12. Drug abuse and medical, psychological or social factors that may interfere with patients' participation in the study or affect the evaluation of the study;
13. Patients have any active autoimmune diseases or a history of autoimmune diseases (including but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, nephritis, hyperthyroidism and decreased thyroid function; patients with vitiligo or with complete remission of asthma in childhood and without any intervention in adulthood may be included; patients with asthma requiring bronchodilators intervention are not included.
14. Received any anti-infection vaccine (e.g. influenza vaccine, chickenpox vaccine, etc.) within 4 weeks before enrollment;
15. Complications require long-term treatment with immunosuppressive drugs, or requiring systemic or local use of immunosuppressive corticosteroids(>10mg/day prednisone or other therapeutic hormones);
16. Any unstable condition or which endangers the patients' safety and compliance;
17. Refuses to sign informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
cCR rate | 3 months after treatment
  cCR rate 3 months after treatment

SECONDARY OUTCOMES:
cCR rate | 6 months after treatment
  cCR rate 6 months after treatment
acute toxicities | from the start of treatment to 3 months after treatment
  acute toxicities
late toxicities | 3 months after treatment
  late toxicities
colostomy rate | from the end of treatment to 2 years after treatment
  colostomy rate
local recurrence rate | from the end of treatment to 5 years after treatment
  local recurrence rate
distant metastasis rate | from the end of treatment to 5 years after treatment
  distant metastasis rate
progression free survival | from the end of treatment to 5 years after treatment
  progression free survival
overall sruvival | from the end of treatment to 5 years after treatment
  overall sruvival

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Study data can be shared after publication of the study results, upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication of study results.

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer Statistics, 2017. CA Cancer J Clin. 2017 Jan;67(1):7-30. doi: 10.3322/caac.21387. Epub 2017 Jan 5. PMID 28055103
- [Background] Amirian ES, Fickey PA Jr, Scheurer ME, Chiao EY. Anal cancer incidence and survival: comparing the greater San-Francisco bay area to other SEER cancer registries. PLoS One. 2013;8(3):e58919. doi: 10.1371/journal.pone.0058919. Epub 2013 Mar 6. PMID 23484057
- [Background] Nigro ND, Vaitkevicius VK, Considine B Jr. Combined therapy for cancer of the anal canal: a preliminary report. 1974. Dis Colon Rectum. 1993 Jul;36(7):709-11. doi: 10.1007/BF02238600. No abstract available. PMID 8348857
- [Background] Epidermoid anal cancer: results from the UKCCCR randomised trial of radiotherapy alone versus radiotherapy, 5-fluorouracil, and mitomycin. UKCCCR Anal Cancer Trial Working Party. UK Co-ordinating Committee on Cancer Research. Lancet. 1996 Oct 19;348(9034):1049-54. PMID 8874455
- [Background] Northover J, Glynne-Jones R, Sebag-Montefiore D, James R, Meadows H, Wan S, Jitlal M, Ledermann J. Chemoradiation for the treatment of epidermoid anal cancer: 13-year follow-up of the first randomised UKCCCR Anal Cancer Trial (ACT I). Br J Cancer. 2010 Mar 30;102(7):1123-8. doi: 10.1038/sj.bjc.6605605. Epub 2010 Mar 16. PMID 20354531
- [Background] Bartelink H, Roelofsen F, Eschwege F, Rougier P, Bosset JF, Gonzalez DG, Peiffert D, van Glabbeke M, Pierart M. Concomitant radiotherapy and chemotherapy is superior to radiotherapy alone in the treatment of locally advanced anal cancer: results of a phase III randomized trial of the European Organization for Research and Treatment of Cancer Radiotherapy and Gastrointestinal Cooperative Groups. J Clin Oncol. 1997 May;15(5):2040-9. doi: 10.1200/JCO.1997.15.5.2040. PMID 9164216
- [Background] Ajani JA, Winter KA, Gunderson LL, Pedersen J, Benson AB 3rd, Thomas CR Jr, Mayer RJ, Haddock MG, Rich TA, Willett C. Fluorouracil, mitomycin, and radiotherapy vs fluorouracil, cisplatin, and radiotherapy for carcinoma of the anal canal: a randomized controlled trial. JAMA. 2008 Apr 23;299(16):1914-21. doi: 10.1001/jama.299.16.1914. PMID 18430910
- [Background] Sana S, Khan AU. Clinical trials in the management of anal cancer. Clin Colon Rectal Surg. 2009 May;22(2):115-9. doi: 10.1055/s-0029-1223843. PMID 20436836
- [Background] Chakravarthy AB, Catalano PJ, Martenson JA, Mondschein JK, Wagner H, Mansour EG, Talamonti MS, Benson AB. Long-term follow-up of a Phase II trial of high-dose radiation with concurrent 5-fluorouracil and cisplatin in patients with anal cancer (ECOG E4292). Int J Radiat Oncol Biol Phys. 2011 Nov 15;81(4):e607-13. doi: 10.1016/j.ijrobp.2011.02.042. Epub 2011 Apr 20. PMID 21514072
- [Background] James RD, Glynne-Jones R, Meadows HM, Cunningham D, Myint AS, Saunders MP, Maughan T, McDonald A, Essapen S, Leslie M, Falk S, Wilson C, Gollins S, Begum R, Ledermann J, Kadalayil L, Sebag-Montefiore D. Mitomycin or cisplatin chemoradiation with or without maintenance chemotherapy for treatment of squamous-cell carcinoma of the anus (ACT II): a randomised, phase 3, open-label, 2 x 2 factorial trial. Lancet Oncol. 2013 May;14(6):516-24. doi: 10.1016/S1470-2045(13)70086-X. Epub 2013 Apr 9. PMID 23578724
- [Background] Olsen JR, Moughan J, Myerson R, Abitbol A, Doncals DE, Johnson D, Schefter TE, Chen Y, Fisher B, Michalski J, Narayan S, Chang A, Crane CH, Kachnic L. Predictors of Radiation Therapy-Related Gastrointestinal Toxicity From Anal Cancer Dose-Painted Intensity Modulated Radiation Therapy: Secondary Analysis of NRG Oncology RTOG 0529. Int J Radiat Oncol Biol Phys. 2017 Jun 1;98(2):400-408. doi: 10.1016/j.ijrobp.2017.02.005. Epub 2017 Feb 13. PMID 28463160
- [Background] Pan YB, Maeda Y, Wilson A, Glynne-Jones R, Vaizey CJ. Late gastrointestinal toxicity after radiotherapy for anal cancer: a systematic literature review. Acta Oncol. 2018 Nov;57(11):1427-1437. doi: 10.1080/0284186X.2018.1503713. Epub 2018 Sep 28. PMID 30264638
- [Background] Hosni A, Han K, Le LW, Ringash J, Brierley J, Wong R, Dinniwell R, Brade A, Dawson LA, Cummings BJ, Krzyzanowska MK, Chen EX, Hedley D, Knox J, Easson AM, Lindsay P, Craig T, Kim J. The ongoing challenge of large anal cancers: prospective long term outcomes of intensity-modulated radiation therapy with concurrent chemotherapy. Oncotarget. 2018 Apr 17;9(29):20439-20450. doi: 10.18632/oncotarget.24926. eCollection 2018 Apr 17. PMID 29755663
- [Background] Russo S, Anker CJ, Abdel-Wahab M, Azad N, Bianchi N, Das P, Dragovic J, Goodman KA, Jones W 3rd, Kennedy T, Kumar R, Lee P, Sharma N, Small W, Suh WW, Jabbour SK. Executive Summary of the American Radium Society Appropriate Use Criteria for Treatment of Anal Cancer. Int J Radiat Oncol Biol Phys. 2019 Nov 1;105(3):591-605. doi: 10.1016/j.ijrobp.2019.06.2544. Epub 2019 Jul 6. No abstract available. PMID 31288054
- [Background] Stewart DB, Gaertner WB, Glasgow SC, Herzig DO, Feingold D, Steele SR; Prepared on Behalf of the Clinical Practice Guidelines Committee of the American Society of Colon and Rectal Surgeons. The American Society of Colon and Rectal Surgeons Clinical Practice Guidelines for Anal Squamous Cell Cancers (Revised 2018). Dis Colon Rectum. 2018 Jul;61(7):755-774. doi: 10.1097/DCR.0000000000001114. No abstract available. PMID 29878949
- [Background] Mullen JT, Rodriguez-Bigas MA, Chang GJ, Barcenas CH, Crane CH, Skibber JM, Feig BW. Results of surgical salvage after failed chemoradiation therapy for epidermoid carcinoma of the anal canal. Ann Surg Oncol. 2007 Feb;14(2):478-83. doi: 10.1245/s10434-006-9221-7. Epub 2006 Nov 14. PMID 17103253
- [Background] Lefevre JH, Parc Y, Kerneis S, Shields C, Touboul E, Chaouat M, Tiret E. Abdomino-perineal resection for anal cancer: impact of a vertical rectus abdominis myocutaneus flap on survival, recurrence, morbidity, and wound healing. Ann Surg. 2009 Nov;250(5):707-11. doi: 10.1097/SLA.0b013e3181bce334. PMID 19801930
- [Background] Ben-Josef E, Moughan J, Ajani JA, Flam M, Gunderson L, Pollock J, Myerson R, Anne R, Rosenthal SA, Willett C. Impact of overall treatment time on survival and local control in patients with anal cancer: a pooled data analysis of Radiation Therapy Oncology Group trials 87-04 and 98-11. J Clin Oncol. 2010 Dec 1;28(34):5061-6. doi: 10.1200/JCO.2010.29.1351. Epub 2010 Oct 18. PMID 20956625
- [Background] Nilsson PJ, Svensson C, Goldman S, Ljungqvist O, Glimelius B. Epidermoid anal cancer: a review of a population-based series of 308 consecutive patients treated according to prospective protocols. Int J Radiat Oncol Biol Phys. 2005 Jan 1;61(1):92-102. doi: 10.1016/j.ijrobp.2004.03.034. PMID 15629599
- [Background] Moureau-Zabotto L, Viret F, Giovaninni M, Lelong B, Bories E, Delpero JR, Pesenti C, Caillol F, de Chaisemartin C, Minsat M, Monges G, Sarran A, Resbeut M. Is neoadjuvant chemotherapy prior to radio-chemotherapy beneficial in T4 anal carcinoma? J Surg Oncol. 2011 Jul 1;104(1):66-71. doi: 10.1002/jso.21866. Epub 2011 Jan 15. PMID 21240983
- [Background] Ott PA, Piha-Paul SA, Munster P, Pishvaian MJ, van Brummelen EMJ, Cohen RB, Gomez-Roca C, Ejadi S, Stein M, Chan E, Simonelli M, Morosky A, Saraf S, Emancipator K, Koshiji M, Bennouna J. Safety and antitumor activity of the anti-PD-1 antibody pembrolizumab in patients with recurrent carcinoma of the anal canal. Ann Oncol. 2017 May 1;28(5):1036-1041. doi: 10.1093/annonc/mdx029. PMID 28453692
- [Background] Shahjehan F, Kamatham S, Ritter A, Kasi PM. Dramatic response to modified docetaxel, cisplatin, and fluorouracil chemotherapy after immunotherapy in a patient with refractory metastatic anal cancer. Clin Case Rep. 2019 Aug 6;7(9):1729-1734. doi: 10.1002/ccr3.2333. eCollection 2019 Sep. PMID 31534737
- [Background] Morris VK, Salem ME, Nimeiri H, Iqbal S, Singh P, Ciombor K, Polite B, Deming D, Chan E, Wade JL, Xiao L, Bekaii-Saab T, Vence L, Blando J, Mahvash A, Foo WC, Ohaji C, Pasia M, Bland G, Ohinata A, Rogers J, Mehdizadeh A, Banks K, Lanman R, Wolff RA, Streicher H, Allison J, Sharma P, Eng C. Nivolumab for previously treated unresectable metastatic anal cancer (NCI9673): a multicentre, single-arm, phase 2 study. Lancet Oncol. 2017 Apr;18(4):446-453. doi: 10.1016/S1470-2045(17)30104-3. Epub 2017 Feb 18. PMID 28223062
- [Background] Rao S, Sclafani F, Eng C, Adams RA, Guren MG, Sebag-Montefiore D, Benson A, Bryant A, Peckitt C, Segelov E, Roy A, Seymour MT, Welch J, Saunders MP, Muirhead R, O'Dwyer P, Bridgewater J, Bhide S, Glynne-Jones R, Arnold D, Cunningham D. International Rare Cancers Initiative Multicenter Randomized Phase II Trial of Cisplatin and Fluorouracil Versus Carboplatin and Paclitaxel in Advanced Anal Cancer: InterAAct. J Clin Oncol. 2020 Aug 1;38(22):2510-2518. doi: 10.1200/JCO.19.03266. Epub 2020 Jun 12. PMID 32530769